CLINICAL TRIAL: NCT00443417
Title: Dose Finding Study to Assess the Efficacy and Safety of SK-PC-B70M in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: A Trial of SK-PC-B70M in Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Clinical research team, SK Chemicals Co.,Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMART_II_2006
Record Dates: First submitted 2007-03-05; First posted 2007-03-06 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2008-01

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — SK-PC-B70M

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 (Placebo Comparator)
  Interventions: Drug: SK-PC-B70M
- 2 (Active Comparator): 200mg qd
  Interventions: Drug: SK-PC-B70M
- 3 (Active Comparator): 200mg bid
  Interventions: Drug: SK-PC-B70M
- 4 (Active Comparator): 400mg qd
  Interventions: Drug: SK-PC-B70M

INTERVENTIONS:
Drug: SK-PC-B70M — dosage, frequency

SUMMARY:
The purpose of this study is to find optimistic dose and to evaluate the efficacy and safety of SK-PC-B70M in patients with mild to moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age range : 50 ~ 85 years
* Clinical diagnosis of probable Alzheimer's disease (DSM-IV and NINCDS-ADRDA criteria)
* MRI within the last 12 months consistent with a diagnosis of AD
* MMSE score 10 to 26
* AChEI or memantine was discontinued at least 3 months prior to screening

Exclusion Criteria:

* Patient in mild cognitive impairment (MCI; CDR-SB <2.5)
* Other central nervous disease
* hypothyroidism, Vitamin B12/ Folic acid deficiency, hypercalcemia, neurosyphilis, AIDS
* T.I.A or Major infarction within the last 12 months
* Any serious disorder that could limit the ability of the patient to participate in the study
* COPD or asthma
* Any condition which would make the patient or the caregiver, in the opinion of the investigator, unsuitable for the study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
ADAS-cog(Alzheimer's Disease Assessment Scale-Cognitive subscale) | 30 minutes

SECONDARY OUTCOMES:
MMSE(Mini Mental State Examination) | 10 minutes
CDR-SB(Clinical Dementia Rating Sum of Box) | 20 minutes
QOL-AD(Quality of Life in Alzheimer's Disease) | 10 minutes
Delayed Word-Recall Task | 5 minute
Symbol Digit Modalities Test | 5 minutes
Digit Backward | 5 minutes
Maze Task | 3 minutes
Digit Cancellation Task | 5 minutes
Verbal Fluency-Categories | 1 minutes
Concentration / Distractibility | 1 minutes
GDS | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Seol Heui Han, MD, PhD, Principal Investigator — Konkuk University Hospital
Locations (1):
- SKchemicalsI nvestigational Site, Seoul, South Korea